CLINICAL TRIAL: NCT01832714
Title: Assessment of Oculomotor, Vestibular and Reaction Time Response Following a Concussive Event
Acronym: NKI-RIF1
Status: Completed | Type: Observational
Sponsor: Neurolign (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NKI-W81XWH-12-C-0205
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Concussion, Mild; Concussion, Intermediate; Concussion, Severe
Keywords: Concussion; mTBI; military; MACE; NKI; NOTC; VNG; VOG; Neuro Kinetics; oculomotor; vestibular; reaction time; I-Portal; eye tracking; Dizziness Handicap Inventory
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mTBI: Subjects who undergo an mTBI event
- Control: Subjects who do not undergo an mTBI

SUMMARY:
This study is designed to evaluate the use of a collection of tests that measure the eye response, balance, oculomotor and reaction time tests to aid in the diagnosis of mTBI. The tests use highly precise measurement tools to assess various neurologic functions. (For example, high-speed cameras to record eye movement, high-end motors to precisely spin and move the subject, comprehensive analysis to stitch together the stimulus and the response.)

Hypotheses:

1. A battery of oculomotor, vestibular and reaction time tests will generate variables that when properly weighted and run through a given multi-variant analysis, will separate the subjects into one of two groups, mTBI or not-mTBI.
2. A battery of neurologic assessment tests including reaction time, vestibular and oculomotor tests taxing a range of neurologic functions and executed using one or more of the I-Portal® family of devices, will generate responses that, when used by a trained physician, can aid in the diagnosis of an mTBI.

DETAILED DESCRIPTION:
The study uses a prospective, between-subjects design comparing an Investigational (mTBI) Group to a Control Group. The Investigational Group includes SM who had been diagnosed with an mTBI. The Control Group consists of SM who do not have clinical symptoms consistent with mTBI. There will be 90 participants in each group, for a target total of 180 study participants

Existing mTBI evaluation tools will be used to qualify the type and severity of a patient's mTBI symptoms. After the volunteer has been assessed by a physician, the following questionnaires and screening tools will be administered:

* Demographic, included control and patient demographics, education, military service, see Appendix A;
* History of health problems and treatments included medication and mTBI history and stress level before testing, including page 1 of MACE, see Appendix B; History of health problems and treatments included medication and mTBI history and stress level before testing, including page 1 of MACE, used for seconds and third tests only, see Appendix B1;
* Glasgow Coma Scale, use only in 24 hrs after accident, see Appendix C;
* Functional Gait Assessment(FGA) - This is an assessment where the individual is asked to perform ten gait tasks. Each gait task is scored by a trained observer on a 0-3 scale (with 0 being could not perform and 3 being performed well). The individual will end up with a total FGA of between 0-30. The test is very sensitive for demonstrating balance dysfunction and improvement.(see Appendix D)
* Trail Making Test (TMT) - This test is a cognitive test in which subjects use a pencil to draw a line between an ordered series of letters or letters/numbers on a paper. Subjects are instructed to follow the appropriate order without lifting the pencil from the paper. Time to completion is a sensitive measure of cognitive performance. (see Appendix E)
* Dizziness Handicap Inventory,(DHI)-This validated questionnaire is commonly used by clinicians to qualify and quantify symptoms associated with dizziness, light-headedness, vertigo, migraine associated dizziness, and to assist with identifying complaints of dizziness related to anxiety, depression, post-traumatic-stress disorder, etc. This tool will capture subjective symptoms associated with mTBI prior to completing the objective measures (see Appendix F)

Device will be comprehensive oculomotor/ neuro-otologic testing system. System components:

* Motorized Chair that can move in up to 3 axis
* Full field Optokinetic stimulus
* Pursuit Tracker™ - laser target generator
* Isolation enclosure
* Patient monitoring and communication technology

FDA classification: The NOTC is covered under an FDA 510K, and certified to standards 60601-1, 60601-1-1, 60601-1-2, and 60601-1-4.

Modifications to approved device:

Included by manufacturer:

1. A new function to existing buttons for reaction time test
2. Audio stimulus for audio reaction time test
3. 2 stationary LED's installed inside enclosure ceiling for crHIT test

Investigational software which incorporates newly defined oculomotor and reaction time tests designed to investigate mTBI will be installed on the device.

ELIGIBILITY:
Inclusion criteria for all subjects (Control and mTBI) - Males or females from 19 - 45years of age and of all races.

Additional Inclusion criteria for mTBI Subjects

- Diagnosed with traumatic brain injury utilizing 2007 DoD Standard diagnosis of

* 1) Exposed to an event,
* 2) Suffered alteration or loss of consciousness secondary to the event, and
* 3) Had a sequelae from the event.

Exclusion criteria for all subjects (Control and mTBI)

* Brain injury resulting from a penetrating wound to the head, neck, face or brain (to include gunshot wounds)
* Presence of severe aphasia
* Persons whom have had an mTBI within the prior month and are symptomatic.
* Persons with a previous history of multiple mTBIs and are symptomatic.
* History of neuropsychiatric disorders antedating the head injury (e.g. hypochondriasis, major depression, schizophrenia)
* Pregnancy
* Prior disorders of hearing and balance including:

  * Meniere's disease
  * Chronic migraine
  * Multiple sclerosis
  * Vestibular neuritis
  * Vestibular schwannoma
  * Sudden sensorineural hearing loss
* Cerebrovascular disorders
* Systemic disorders: e.g. chronic renal failure, cirrhosis of the liver, etc.
* Medications which depress the sensorium precluding patient compliance with the testing (considered on a case-by-case basis)
* Previous contraindicating surgeries at the discretion of the study physicians or audiologists

Additional Exclusion criteria for Control Subjects

* Concussion within the last year (12 months)
* Repeated blast exposure

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Investigational Group includes Service Members (SM) and civilians who had been diagnosed with an mTBI. The Control Group consists of SM and civilians who do not have clinical symptoms consistent with mTBI. There will be at least 90 participants in each group, for a target total of at least 180 study participants.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Variability of latency in reflexive saccades (ms) | within 7 days of a concussion event
  Examine the latency of subjects with mTBI with respect to mean latency and standard deviation of control subjects.
Variability of latency in reaction time test (ms) | within 7 days of a concussion event
  Examine the latency of subjects with mTBI with respect to mean latency and standard deviation of control subjects.
Variability of error in subjective visual vertical test (degrees) | within 7 days of a concussion event
  Examine the mean error of subjects with mTBI with respect to mean error and standard deviation of control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Kiderman, PhD ME, Principal Investigator — Neuro Kinetics, Inc
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Madigan Army Medical Center, Tacoma, Washington